CLINICAL TRIAL: NCT01650467
Title: Imatinib Response in Patients With Chronic Myeloid Leukemia (CML) in Function of Abl Polymorphisms
Acronym: abl LMC
Status: Withdrawn | Type: Observational
Why Stopped: Funding is late, unforseeable.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2012/JBG-02; 2012-A00639-34 (Other: RCB number)
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Leukemia, Myeloid, Chronic-Phase
Keywords: abl polymorphisms
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Two 7 ml EDTA tubes for genotyping abl and bcr-abl polymorphisms
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy controls: 60 healthy controls with no hematological pathologies
- Imatinib optimal response: 30 CML patients who are optimal responders to imatinib treatment
- Imatinib primary resistance: 30 CML patients who have primary resistance to imatinib treatment

SUMMARY:
The main objective of this study is to evaluate the existence of a relationship between the presence of certain abl polymorphisms (or haplotypes) upon CML diagnosis and the occurrence of primary resistance to the treatment of CML by imatinib.

DETAILED DESCRIPTION:
The first secondary objective of this study is to identify, in patients not responding to treatment, possible changes in the polymorphisms of interest during the course of the disease, reclassifying such polymorphisms as mutations.

The second secondary objective is to compare the control patients in terms of polymorphism frequency on the nonpathological abl fraction.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan

Inclusion Criteria for all CML patients

* Patients diagnosed with CML
* Treatment with Imatinib in first-line monotherapy and this for at least 12 months
* RNA and / or cDNA used for diagnosis correctly stored in the biobank

Inclusion Criteria for CML patients already having undergone a follow-up visit at 12 months

* RNA and / or cDNA used for diagnosis/follow-up correctly stored in the biobank
* Cytogenetic results are available
* Absence of ITK mutation for the primary resistance subgroup
* Validated compliance

Inclusion Criteria for the optimal response group:

* bcr-abl typing is less than 0.1% at 12 months

Inclusion criteria for the primary resistance group

* bcr-abl typings is >1% and/or Philadelphia+ is greater than 0

Inclusion Criteria for the control population

* Absence of hematologic malignancy

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient has a contraindication for a treatment used in this study

Exclusion Criteria for CML patients already having undergone a follow-up visit at 12 months

* Known or suspected cause for resistance (dose reduced due to intolerance, digestive disease responsible for malabsorption ...)

Exclusion Criteria for the control population

* History or suspicion of hemopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will include 60 healthy controls (free of hematologic pathology, seen in genetic counseling) and stratify the recruitment of patients with CML among 30 patients with optimal imatinib response and 30 with primary resistance.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
abl genotype | baseline ; at diagnosis
  The abl genotype will be determined for all subjects

SECONDARY OUTCOMES:
abl genotype | 12 months after diagnosis
  The abl genotype will be determined for all subjects
bcr-abl leucemic fraction genotype | 12 months after diagnosis
  The bcr-able leucemic fraction genotype will be determined for CML patients
bcr-abl leucemic fraction genotype | baseline ; at diagnosis
  The bcr-able leucemic fraction genotype will be determined for CML patients
abl non-leucemic fraction genotype | baseline ; at diagnosis
  The abl non-leucemic fraction genotype will be determined for CML patients
abl non-leucemic fraction genotype | 12 months after diagnosis
  The abl non-leucemic fraction genotype will be determined for CML patients

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Gaillard, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (3):
- France (3):
  - Clinique du Parc, Castelnau-le-Lez
  - CHU de Montpellier - Hôpital Saint-Eloi, Montpellier
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes